CLINICAL TRIAL: NCT00416598
Title: Phase II Study of Maintenance Therapy With Decitabine (NSC #127716) Following Standard Induction and Cytogenetic Risk-Adapted Intensification in Previously Untreated Patients With AML < 60 Years
Brief Title: Decitabine as Maintenance Therapy After Standard Therapy in Treating Patients With Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00444; NCI-2009-00444 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000521603; CALGB 10503 (Other: Alliance for Clinical Trials in Oncology); CALGB-10503 (Other: CTEP); R21CA128377 (NIH); U10CA180821 (NIH); U10CA031946 (NIH); NCT01647074 (obsolete NCT alias)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22.3;q23.3); MLLT3-KMT2A; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute | interventions — Busulfan; Cytarabine; Daunorubicin; Decitabine; Injections; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (1):
- Treatment (chemotherapy, PBSC or bone marrow transplantation) (Experimental): See Detailed Description.
  Interventions: Procedure: Autologous Bone Marrow Transplantation; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Decitabine; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Procedure: Autologous Bone Marrow Transplantation — Undergo autologous bone marrow transplantation
  Other Names: ABMT; Autologous Bone Marrow Transplant; Autologous Marrow Transplantation
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSC transplantation
  Other Names: Autologous Hematopoietic Cell Transplantation; autologous stem cell transplantation
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Aza-TdC; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well decitabine works when given as maintenance therapy after standard therapy in treating patients with previously untreated acute myeloid leukemia. Drugs used in chemotherapy, such as cytarabine, daunorubicin, etoposide, busulfan, and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving decitabine as maintenance therapy after standard therapy may keep cancer cells from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy, feasibility, and toxicities when one year of maintenance therapy with decitabine is given to patients < 60 years with untreated acute myeloid leukemia (AML) who achieve and maintain first complete remission (CR) following an established induction and intensification regimen.

II. To determine the 1-year disease free survival rate for AML patients in first CR treated with maintenance decitabine.

SECONDARY OBJECTIVES:

I. To measure biologic response to decitabine in evaluable patients with fusion genes to determine eradication of minimal residual disease.

II. To measure surrogates for deoxyribonucleic acid (DNA) demethylation including downregulation of DNA methyltransferase 1 (DNMT1) and induction of fetal hemoglobin.

III. To examine the significance of gene re expression following ex vivo decitabine exposure in primary AML cells taken at the time of diagnosis on clinical outcome and on gene expression at the time of relapse after in vivo decitabine exposure.

IV. To continue to evaluate the effectiveness of a cytogenetically risk-adapted approach for consolidation therapy for patients with core binding factor (CBF) or non-CBF AML.

V. To continue the investigation begun in Cancer and Leukemia Group B (CALGB) 19808 aimed at correlation of the rate of relapse and toxicity with intravenous (IV) busulfan pharmacokinetics when busulfan and etoposide are used as the preparative regimen for autologous stem cell transplantation for AML patients in first CR.

VI. To correlate outcome measures such as complete response (CR), disease-free survival (DFS), event-free survival (EFS), and overall survival (OS), with pretreatment characteristics such as age, sex, race, blood counts, morphology, immunophenotype, cytogenetics, and molecular features of AML.

OUTLINE:

REMISSION INDUCTION THERAPY: Patients receive cytarabine IV over 168 hours on days 1-7 and daunorubicin hydrochloride IV over 5-10 minutes and etoposide IV over 2 hours on days 1-3. Patients undergo bone marrow biopsy on day 14. Patients with residual leukemia proceed to second remission induction therapy. Patients achieving complete remission (CR) proceed to intensification therapy.

SECOND REMISSION INDUCTION THERAPY: Patients receive cytarabine IV over 120 hours on days 1-5 and daunorubicin hydrochloride IV and etoposide IV over 2 hours on days 1 and 2. Patients undergo bone marrow biopsy on day 42. Patients with residual leukemia are removed from the study. Patients achieving CR proceed to intensification therapy.

INTENSIFICATION THERAPY: Patients are stratified and receive intensification therapy according to cytogenetic findings (favorable cytogenetics [t(8;21)(q22q22), inv(16)(p13;q22), or t(16;16)(p13;q22) by cytogenetic and/or molecular analysis] vs unfavorable cytogenetics [all other cytogenetic findings, including normal cytogenetics]).

FAVORABLE CYTOGENETICS: Within 2-4 weeks after achieving CR, patients receive high-dose cytarabine IV over 3 hours twice daily on days 1, 3, and 5.

Treatment repeats every 28 days for up to 3 courses.

UNFAVORABLE CYTOGENETICS: Peripheral blood stem cell (PBSC) mobilization: Within 2-4 weeks after achieving CR, patients receive etoposide IV over 96 hours and high-dose cytarabine IV over 2 hours twice daily on days 1-4 and filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 14 and continuing until blood counts recover. Patients then proceed to transplantation.

PBSC OR BONE MARROW TRANSPLANTATION: Patients receive busulfan IV over 2 hours 4 times daily on days -7 to -4 and etoposide IV over 4 hours on day -3. Patients undergo autologous PBSC or bone marrow transplantation on day 0 and receive G-CSF SC once daily beginning on day 0 and continuing until blood counts recover.

UNFAVORABLE CYTOGENETICS AND UNABLE TO UNDERGO PBSC TRANSPLANTATION: Within 2-4 weeks after achieving CR, patients receive etoposide, high-dose cytarabine, and G-CSF as in unfavorable cytogenetics (PBSC mobilization) followed by 2 courses of high-dose cytarabine as in favorable genetics.

MAINTENANCE THERAPY: Within 60-90 days after completion of intensification therapy, patients receive decitabine IV over 1 hour on days 1-5. Treatment repeats every 6 weeks for up to 8 courses.

After completion of study treatment, patients are followed up every 2 months for 1 year, every 6 months for 2 years, and then yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal histologic diagnosis of AML (> 20% blasts in the bone marrow based on the World Health Organization [WHO] and/or French American British [FAB] classifications), excluding M3 (acute promyelocytic leukemia); patients with antecedent myelodysplasia are eligible for treatment on this trial only if there were no bone marrow biopsy showing myelodysplastic syndrome (MDS) > 3 months prior to enrollment; patients with therapy-related AML are eligible if they have been free of their primary disease and have not received any chemotherapy for at least 2 years
* No prior 5-azacitidine or decitabine therapy
* No prior treatment for leukemia or myelodysplastic syndrome with four permissible exceptions:

  * Emergency leukapheresis
  * Emergency treatment for hyperleukocytosis with hydroxyurea
  * Cranial radiation therapy (RT) for central nervous system (CNS) leukostasis (one dose only)
  * Growth factor/cytokine support

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 546 (Actual)
Dates: Start 2006-11-15 (Actual); Primary Completion 2011-01-31 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Blum, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (46):
- United States (46):
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Florida Hospital Orlando, Orlando, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - Veterans Administration, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont

REFERENCES:
- [Derived] Seffernick AE, Mrozek K, Nicolet D, Stone RM, Eisfeld AK, Byrd JC, Archer KJ. High-dimensional genomic feature selection with the ordered stereotype logit model. Brief Bioinform. 2022 Nov 19;23(6):bbac414. doi: 10.1093/bib/bbac414. PMID 36184192
- [Derived] Yin J, LaPlant B, Uy GL, Marcucci G, Blum W, Larson RA, Stone RM, Mandrekar SJ. Evaluation of event-free survival as a robust end point in untreated acute myeloid leukemia (Alliance A151614). Blood Adv. 2019 Jun 11;3(11):1714-1721. doi: 10.1182/bloodadvances.2018026112. PMID 31171508
- [Derived] Blum W, Sanford BL, Klisovic R, DeAngelo DJ, Uy G, Powell BL, Stock W, Baer MR, Kolitz JE, Wang ES, Hoke E, Mrozek K, Kohlschmidt J, Bloomfield CD, Geyer S, Marcucci G, Stone RM, Larson RA; Alliance for Clinical Trials in Oncology. Maintenance therapy with decitabine in younger adults with acute myeloid leukemia in first remission: a phase 2 Cancer and Leukemia Group B Study (CALGB 10503). Leukemia. 2017 Jan;31(1):34-39. doi: 10.1038/leu.2016.252. Epub 2016 Sep 13. PMID 27624549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2006 and July 2010, 546 participants were recruited.
Groups:
- Treatment (Chemotherapy, PBSC or Bone Marrow Transplantation): See Detailed Description:
  Patients undergo induction therapy comprising cytarabine and daunorubicin hydrochloride. Patient with RD undergo second induction therapy comprising cytarabine, daunorubicin hydrochloride, and etoposide. Patients with CR and favorable cytogenetics who achieve CR receive intensification therapy comprising high-dose cytarabine. Patients with UC receive etoposide, high-dose cytarabine, G-CSF., and busulfan and proceed to PBSC or bone marrow transplantation. Patients with UC and unable to undergo transplantation receive etoposide, high-dose cytarabine, and G-CSF. Patients then receive decitabine as maintenance therapy.
Period: Induction & Intensification
Arm/Group | Treatment (Chemotherapy, PBSC or Bone Marrow Transplantation)
Started | 546
Completed | 134
Not Completed | 412
Not completed — Adverse Event | 38
Not completed — Death | 32
Not completed — Withdrawal by Subject | 46
Not completed — Alternative Treatment | 135
Not completed — Physician discretion/other medical issue | 45
Not completed — Relapse/progression | 29
Not completed — Failed induction | 87
Period: Decitabine Maintenance
Arm/Group | Treatment (Chemotherapy, PBSC or Bone Marrow Transplantation)
Started | 134
Completed | 62
Not Completed | 72
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 18
Not completed — Progression/relapse | 38
Not completed — Alternative treatment | 2
Not completed — Physician discretion/other medical issue | 9

BASELINE CHARACTERISTICS:
Population: Participants who received investigational decatibine maitenance were analyzed.
Groups:
- Decatibine Maintenance: Within 60-90 days after completion of intensification therapy, patients receive 20 mg/m^2 decitabine IV over 1 hour on days 1-5. Treatment repeats every 6 weeks for up to 8 courses.
Arm/Group | Decatibine Maintenance
Number analyzed (Participants) | 134
Age, Continuous [Median (Full Range); unit: years] | 45 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 111
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Maintenance Decitabine.
Description: To determine feasibility of decitabine maintenance, this outcome measures the number of participants who completed all 8 planned cycles of decitabine maintenance as per protocol.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Decatibine Maintenance
Number analyzed (Participants) | 134
participants | 62

2. Primary Outcome: Disease-free Survival (DFS) Rate at 1 Year
Description: For participants who achieved a complete remission (CR), this is the percentage of participants who were alive and relapse free at 1 year. The 1 year rate, with 95% confidence interval, was estimated using the Kaplan-Meier method
  A CR is defined as those with > 20% cellularity of bone marrow biopsy, no presence of extramedullary leukemia for AML, <5 % myeloblast cells for bone marrow with peripheral blood and normal complete blood count (absolute neutrophils > 1000 mL and platelets >= 100,000 mL).
Time Frame: At 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Decatibine Maintenance
Number analyzed (Participants) | 134
percentage of participants | 80

3. Other Pre Specified Outcome: Relationship Between Busulfan Pharmacokinetics (Area Under the Curve) and Relapsed Disease
Description: Results from busulfan pharmacokinetics will be pooled with those from CALGB 19808.
Time Frame: At baseline, after 2, 4, and 6 hours after the start of busulfan infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: 132 participants were assessed for adverse events during decitabine maintenance
Arm/Group | Decatibine Maintenance
Serious Adverse Events (participants affected / at risk) | 0/132
Other Adverse Events (participants affected / at risk) | 130/132
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decatibine Maintenance (N=132)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (18)
Hemoglobin decreased (Blood and lymphatic system disorders) | 125 (488)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (5)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Cardiac pain (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 5 (7)
Palpitations (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 11 (16)
Ear disorder (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 4 (7)
Hypothyroidism (Endocrine disorders) | 1 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 2 (2)
Eye disorder (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Flashing vision (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 6 (7)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 21 (25)
Anal exam abnormal (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 30 (52)
Diarrhea (Gastrointestinal disorders) | 28 (47)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 5 (9)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 5 (5)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 4 (5)
Hemorrhoids (Gastrointestinal disorders) | 5 (6)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 64 (161)
Oral pain (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Salivary gland disorder (Gastrointestinal disorders) | 1 (2)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 3 (4)
Tooth disorder (Gastrointestinal disorders) | 2 (5)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 26 (41)
Chest pain (General disorders) | 7 (7)
Chills (General disorders) | 16 (19)
Edema limbs (General disorders) | 16 (28)
Fatigue (General disorders) | 89 (283)
Fever (General disorders) | 15 (16)
Flu-like symptoms (General disorders) | 2 (3)
General symptom (General disorders) | 3 (3)
Ill-defined disorder (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 20 (26)
Visceral edema (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (3)
Hepatobiliary disease (Hepatobiliary disorders) | 2 (2)
Autoimmune disorder (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Immune system disorder (Immune system disorders) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5)
Catheter related infection (Infections and infestations) | 7 (9)
Conjunctivitis infective (Infections and infestations) | 2 (2)
Gingival infection (Infections and infestations) | 3 (6)
Infection (Infections and infestations) | 10 (13)
Lip infection (Infections and infestations) | 2 (2)
Mucosal infection (Infections and infestations) | 2 (2)
Opportunistic infection (Infections and infestations) | 2 (3)
Otitis media (Infections and infestations) | 3 (4)
Peripheral nerve infection (Infections and infestations) | 2 (4)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 10 (10)
Skin infection (Infections and infestations) | 3 (3)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 15 (17)
Ureteritis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (6)
Vaginal infection (Infections and infestations) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 5 (7)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 57 (159)
Alkaline phosphatase increased (Investigations) | 26 (74)
Aspartate aminotransferase increased (Investigations) | 49 (110)
Blood bilirubin increased (Investigations) | 16 (20)
Creatinine increased (Investigations) | 11 (19)
Gamma-glutamyltransferase increased (Investigations) | 2 (6)
INR increased (Investigations) | 4 (5)
Laboratory test abnormal (Investigations) | 14 (26)
Leukocyte count decreased (Investigations) | 60 (257)
Lymphocyte count decreased (Investigations) | 41 (147)
Neutrophil count decreased (Investigations) | 127 (609)
Platelet count decreased (Investigations) | 127 (604)
Serum cholesterol increased (Investigations) | 1 (3)
Weight gain (Investigations) | 7 (21)
Weight loss (Investigations) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 19 (33)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 5 (12)
Blood glucose increased (Metabolism and nutrition disorders) | 57 (149)
Blood uric acid increased (Metabolism and nutrition disorders) | 6 (22)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 17 (27)
Serum calcium decreased (Metabolism and nutrition disorders) | 21 (33)
Serum calcium increased (Metabolism and nutrition disorders) | 4 (4)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (6)
Serum magnesium decreased (Metabolism and nutrition disorders) | 9 (22)
Serum phosphate decreased (Metabolism and nutrition disorders) | 8 (22)
Serum potassium decreased (Metabolism and nutrition disorders) | 22 (38)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 18 (29)
Serum sodium increased (Metabolism and nutrition disorders) | 3 (4)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (38)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (71)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (21)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (38)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (9)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (45)
Abducens nerve disorder (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 25 (39)
Dysgeusia (Nervous system disorders) | 7 (12)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 39 (71)
Memory impairment (Nervous system disorders) | 4 (10)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 4 (5)
Peripheral motor neuropathy (Nervous system disorders) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 28 (63)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 3 (3)
Speech disorder (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 31 (57)
Confusion (Psychiatric disorders) | 4 (9)
Depression (Psychiatric disorders) | 19 (43)
Insomnia (Psychiatric disorders) | 26 (59)
Libido decreased (Psychiatric disorders) | 2 (2)
Personality change (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 2 (2)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (4)
Kidney pain (Renal and urinary disorders) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 5 (6)
Urogenital disorder (Renal and urinary disorders) | 3 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 2 (4)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 1 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 8 (13)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 17 (31)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (68)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 (49)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (16)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (14)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 17 (30)
Skin disorder (Skin and subcutaneous tissue disorders) | 12 (20)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 12 (14)
Flushing (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 14 (24)
Hypotension (Vascular disorders) | 8 (8)
Thrombosis (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less